CLINICAL TRIAL: NCT04630951
Title: Effects of Blood Flow Restriction Resistance Training on Muscle Characteristics, Strength and Performance of Professional Soccer Players
Brief Title: Blood Flow Restriction Strength Training in Professional Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160CER20
Record Dates: First submitted 2020-10-28; First posted 2020-11-16 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Resistance Training; Blood Pressure
Keywords: Strenght Training; Soccer; Blood Flood Restriction; Performance; Sport Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength training based on low loads with blood flow restriction (Experimental group I) (Experimental): 1. Squat
  2. Single Deadlift
  3. Back Squat
  Interventions: Other: Blood Flow Restriction Strength training with low load
- Strenght training based on high loads (Experimental group II) (Experimental): 1. Squat
  2. Single Deadlift
  3. Back Squat
  Interventions: Other: High Load Strength Training

INTERVENTIONS:
Other: Blood Flow Restriction Strength training with low load — Low Load (20-50% 1RM), 4 set of 30/15/15/15 repetitions, 30 seconds resting between sets.
  Arms: Strength training based on low loads with blood flow restriction (Experimental group I)
Other: High Load Strength Training — High Load (60-80% 1RM) 4 sets of 8 repetitions, 2 minutes resting between sets
  Arms: Strenght training based on high loads (Experimental group II)

SUMMARY:
The aims of this clinical study are evaluated the effects of Blood Flood Restriction training on the sport performance of professional and semi-professional soccer players. The participants are twenty male professional and semi-professional soccer players who are playing at RCD Mallorca. Participants will be assigned in two different groups. Both groups develop for six weeks a strength training programs. The first group will base their training in Low Load using Blood Flow Restriction (20-50% of one maximum repetition). The second group will base their training in High Load (60-80% of one maximum repetition). This training program includes three type of exercises in each training session; back squat, single deadlift and barbell hip thrust. Before and after this program the investigators will collect sociodemographic and anthropometrics data. On top of that, the investigators will evaluate the muscle mass, the electrical activity produced by skeletal muscles, the muscle strength and the sprint ability of every participant. Before to the evaluation, the soccer players will warm-up during 15 minutes under the control of the evaluators.

DETAILED DESCRIPTION:
PARTICIPANTS:

Participants are soccer players of RCD Mallorca (Second Spanish Football Division) and RCD Mallorca B (Third Spanish Football Division).Before to start the study, every participant will receive an informed consent about the clinical study. This informed consent will be signed by them according to Declaration of Helsinki. At the same time, the data will be anonymized and only the main researcher of the study will have access to it, to ensure compliance with the Data Protection Law.

W-UP:

The warm-up will consist of 5 minutes running slow (treadmill), 5 minutes mobility, and 5 minutes of running exercises. In addition, the warm-up will contain a familiarization with the jump test

ELIGIBILITY:
Inclusion Criteria:

* No injuries in the last 6 months
* 1 years experience minimun in the division.

Exclusion Criteria:

* Amateurs players

Ages: 14 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Muscle Mass | Change from Baseline in Muscle Mass at 6 Weeks
  Muscle Mass mesured with measuring tape
Change from Baseline in Maximum Voluntary Isometric Contraction (MVIC) | Change from Baseline in Maximum voluntary Isometric Contraction at 6 Weeks
  MVIC mesured by Force Platform (Vald Performance, Brisbane, QLD)
Change from Baseline in Electrical Muscle Activity | Change from Baseline in Electrical Muscle Activity at 6 weeks
  Electrical Muscle Activity mesured by Surface Electromyography (mDurance®, España)
Change from Baseline in Countermovement Jump (CMJ) | Change from Baseline in countermovement Jump (CMJ Test) at 6 weeks
  CMJ Test measured by Force Platform (Vald Performance, Brisbane, QLD)
Change from in Force-Velocity Profile (F-V) | Change from Baseline in Force-Velocity Profile at 6 Weeks
  F-V Profile measured by MyJump App
Change from Baseline in Sprint Ability | Change from Baseline in Sprint Ability at 6 weeks
  Sprint Ability measured by MySprint App
Change from Post-Intervention in Sport Injuries Incidence | Change from Post-Intervention up to 8 months.
  Incidence of injuries related to sport practice

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Romero Franco, Study Director — University of Balearic Islands; Christian Castilla López, Principal Investigator — University of Balearic Islands
Locations (1):
- Christian, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No